CLINICAL TRIAL: NCT06498440
Title: Comparative Efficacy of NSAID and Steroid-NSAID Combination Following Selective Laser Trabeculoplasty: a Phase 4, Single-centre, Randomized Controlled Trial
Brief Title: Efficacy of NSAID vs. Steroid-NSAID Combo Post-Selective Laser Trabeculoplasty: Phase 4, Single-Center RCT
Acronym: CES-NSLT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Enitan Sogbesan, Dr. Enitan Sogbesan, Principal Investigator, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 17189
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension; Postoperative Inflammation
Keywords: Selective Laser Trabeculoplasty (SLT); Non-steroidal anti-inflammatory drugs (NSAIDs); Ketorolac; Fluorometholone; Postoperative care; Intraocular pressure (IOP); Visual acuity; Glaucoma treatment; Ophthalmology; Randomized controlled trial (RCT)
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Ketorolac; Ophthalmic Solutions; Ketorolac Tromethamine; Fluorometholone

STUDY DESIGN:
Intervention Model Description: This study is a Phase 4 single-centre randomized controlled trial (RCT) at the Hamilton Regional Eye Clinic, St. Joseph's Healthcare Hamilton. It aims to compare postoperative treatments following Selective Laser Trabeculoplasty (SLT) in open-angle glaucoma patients. Participants are randomly assigned to one of three groups: ketorolac alone, ketorolac with fluorometholone, or no treatment (control). The primary outcome is the change in intraocular pressure (IOP) from baseline to one year post-SLT, with secondary outcomes including visual acuity, inflammation, and patient-reported discomfort. Follow-up assessments occur at 1 hour, 1 week, 1 month, 3 months, 6 months, and 1 year. The study follows CONSORT guidelines and has ethical approval from the Hamilton Integrated Research Ethics Board (HiREB). The goal is to provide reliable data on effective postoperative management strategies, enhancing clinical practice in glaucoma treatment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Ketorolac Alone (Experimental): Participants in this arm will receive ketorolac 0.5% eye drops administered twice daily for one week following Selective Laser Trabeculoplasty (SLT). Ketorolac is a non-steroidal anti-inflammatory drug (NSAID) that helps reduce inflammation and alleviate pain. The purpose of this intervention is to assess the efficacy and safety of ketorolac alone in managing postoperative inflammation and patient comfort compared to other treatment strategies.
  Interventions: Drug: Ketorolac 0.5% Eye Drops
- Ketorolac with Fluorometholone (Experimental): Participants in this arm will receive a combination of ketorolac 0.5% eye drops administered twice daily and fluorometholone 0.1% eye drops administered four times daily for one week following Selective Laser Trabeculoplasty (SLT). Fluorometholone is a corticosteroid that reduces inflammation by stabilizing capillary permeability and inhibiting inflammatory cell activation. This arm aims to evaluate the combined efficacy and safety of ketorolac and fluorometholone in postoperative care.
  Interventions: Drug: Ketorolac 0.5% and Fluorometholone 0.1% Eye Drops
- No Treatment Control (No Intervention): Participants in this arm will not receive any postoperative treatment following Selective Laser Trabeculoplasty (SLT). This control group is included to provide a baseline for comparison against the treatment groups receiving ketorolac alone or a combination of ketorolac and fluorometholone. The purpose is to assess the natural course of postoperative inflammation and patient comfort without intervention.

INTERVENTIONS:
Drug: Ketorolac 0.5% Eye Drops — Participants in this arm will receive ketorolac 0.5% eye drops, administered twice daily for one week following Selective Laser Trabeculoplasty (SLT). Ketorolac is a non-steroidal anti-inflammatory drug (NSAID) that works by inhibiting cyclooxygenase (COX) enzymes, which play a key role in the inflammatory process. This intervention aims to reduce postoperative inflammation and pain, promoting patient comfort and potentially improving outcomes following SLT.
  Other Names: Acular; Acular LS; Acuvail
  Arms: Ketorolac Alone
Drug: Ketorolac 0.5% and Fluorometholone 0.1% Eye Drops — Participants in this arm will receive a combination of ketorolac 0.5% eye drops and fluorometholone 0.1% eye drops. Ketorolac will be administered twice daily and fluorometholone four times daily for one week following SLT. Fluorometholone is a corticosteroid that reduces inflammation by stabilizing capillary permeability and inhibiting inflammatory cell activation. The combination aims to maximize anti-inflammatory effects and enhance patient comfort, potentially leading to better postoperative outcomes compared to ketorolac alone or no treatment.
  Other Names: FML; Acular; Acuvail; Fluor-Op
  Arms: Ketorolac with Fluorometholone

SUMMARY:
This clinical trial, led by Dr. Enitan A. Sogbesan at the Hamilton Regional Eye Clinic, St. Joseph's Healthcare Hamilton, aims to compare the efficacy and safety of non-steroidal anti-inflammatory drug (NSAID) ketorolac alone versus a combination of ketorolac and the corticosteroid fluorometholone, and a control group receiving no postoperative treatment. The trial will evaluate these treatment strategies following Selective Laser Trabeculoplasty (SLT) in patients with open-angle glaucoma. The primary objective is to determine the most effective postoperative management strategy to reduce inflammation, improve patient comfort, and control intraocular pressure (IOP). Participants will be randomly assigned to one of the three groups, with follow-up visits scheduled at 1 hour, 1 week, 1 month, 3 months, 6 months, and 1 year post-SLT. The study's findings aim to guide clinicians in optimizing postoperative care for better patient outcomes.

DETAILED DESCRIPTION:
Selective Laser Trabeculoplasty (SLT) is a widely used procedure introduced by Latina and Park in 1995 for the management of various forms of glaucoma, including open-angle glaucoma (OAG), pigmentary glaucoma, pseudoexfoliation glaucoma, and ocular hypertension. SLT helps prevent irreversible blindness by effectively managing these conditions. However, postoperative management strategies vary among practitioners, with some prescribing NSAIDs, a combination of NSAIDs and steroids, or no treatment at all. There is no consensus on the most effective and safest approach.

This phase 4 single-centre randomized controlled trial seeks to address this knowledge gap by comparing the postoperative effects of ketorolac alone, a combination of ketorolac and fluorometholone, and a no treatment control group on inflammation and patient comfort following SLT. The hypothesis is that treatment with ketorolac alone or in combination with fluorometholone will show superior results in reducing inflammation and improving patient comfort compared to no treatment.

The study will enroll patients undergoing SLT at the Hamilton Regional Eye Clinic. Participants will be randomized into either one of two treatment groups or one control group (no treatment) and monitored for changes in IOP, visual acuity, patient comfort, and the occurrence of any complications over a one-year period. Data collected from these assessments will be analyzed to determine the comparative efficacy and safety of the three strategies.

Inclusion criteria include adults diagnosed with open-angle glaucoma, IOP greater than 16 mmHg, and visual acuity of 20/200 or better. Exclusion criteria include recent ocular surgeries, allergies to ketorolac or fluorometholone, and pregnancy. The primary outcome measure is the change in IOP from baseline, while secondary outcomes include visual acuity, anterior chamber inflammation, and patient-reported discomfort.

The trial follows CONSORT guidelines to maintain transparency and reproducibility. Ethical approval will be obtained from the Hamilton Integrated Research Ethics Board (HiREB), ensuring compliance with ethical and legal requirements.

The results of this study will inform postoperative care decisions following SLT, potentially leading to improved patient outcomes and satisfaction. This trial also aims to contribute to a more standardized postoperative management protocol for SLT, enhancing clinical practice and patient care in glaucoma treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older.
* Diagnosed with open-angle glaucoma.
* Intraocular pressure (IOP) greater than 16 mmHg on at least two consecutive occasions separated by one month.
* Visual acuity of 20/200 or better in at least one eye.
* Provided informed consent.

Exclusion Criteria:

* Patients with any other ocular disorders or surgeries within the last six months.
* Allergy or intolerance to ketorolac or fluorometholone.
* Previous use of systemic ketorolac or fluorometholone in the past month.
* Pregnancy or breastfeeding.
* Patients who are unable to speak/understand English.
* Any condition that in the investigator's opinion would make participation not in the best interest of the patient or could prevent, limit, or confound the protocol-specified assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Intraocular Pressure (IOP) from Baseline | Baseline to 1 year post-SLT
  The primary outcome measure is the mean change in intraocular pressure (IOP) from baseline to 1 year post-Selective Laser Trabeculoplasty (SLT). IOP will be measured using Goldmann applanation tonometry (GAT) at each follow-up visit. The baseline IOP is determined as the average of measurements taken on the day of SLT booking and on the day of the SLT procedure. The primary objective is to compare the effectiveness of ketorolac alone, ketorolac with fluorometholone, and no treatment in reducing IOP following SLT.

SECONDARY OUTCOMES:
Visual Acuity | Baseline to 1 year post-SLT
  Visual acuity will be measured using a Snellen chart and reported in logMAR units at each follow-up visit. The study will compare changes in visual acuity among the three treatment groups to determine the impact of each postoperative strategy on visual function.
Anterior Chamber Inflammation | Baseline to 1 year post-SLT
  Anterior chamber inflammation will be assessed using the Standardization of Uveitis Nomenclature (SUN) Working Group grading system. The presence and severity of cells and flare in the anterior chamber will be evaluated at each follow-up visit to compare the anti-inflammatory effects of the treatment strategies.
Patient-Reported Discomfort | Baseline to 1 year post-SLT
  Patient discomfort will be recorded at each follow-up visit. Participants will rate their discomfort on a scale, allowing for comparison of patient comfort levels across the three treatment groups.
Incidence of Postoperative Complications | Baseline to 1 year post-SLT
  The incidence of postoperative complications, such as ocular discomfort, conjunctival hyperemia, and corneal abrasions, will be recorded at each follow-up visit. This measure will help determine the safety profile of ketorolac alone, ketorolac with fluorometholone, and no treatment following SLT.

CONTACTS AND LOCATIONS:
Overall Officials: Enitan A Sogbesan, MD, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton Regional Eye Institute, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The decision to share individual participant data (IPD) with other researchers is currently under consideration. The final decision will be made in alignment with institutional policies and ethical guidelines to ensure the protection of participant confidentiality and the integrity of the study.

REFERENCES:
- [Background] Canadian Ophthalmological Society Glaucoma Clinical Practice Guideline Expert Committee; Canadian Ophthalmological Society. Canadian Ophthalmological Society evidence-based clinical practice guidelines for the management of glaucoma in the adult eye. Can J Ophthalmol. 2009;44 Suppl 1:S7-93. doi: 10.3129/cjo44s1. No abstract available. English, French. PMID 19492005
- [Background] Foster PJ, Buhrmann R, Quigley HA, Johnson GJ. The definition and classification of glaucoma in prevalence surveys. Br J Ophthalmol. 2002 Feb;86(2):238-42. doi: 10.1136/bjo.86.2.238. PMID 11815354
- [Background] Zhang N, Wang J, Li Y, Jiang B. Prevalence of primary open angle glaucoma in the last 20 years: a meta-analysis and systematic review. Sci Rep. 2021 Jul 2;11(1):13762. doi: 10.1038/s41598-021-92971-w. PMID 34215769
- [Background] Farkouh A, Frigo P, Czejka M. Systemic side effects of eye drops: a pharmacokinetic perspective. Clin Ophthalmol. 2016 Dec 7;10:2433-2441. doi: 10.2147/OPTH.S118409. eCollection 2016. PMID 27994437
- [Background] Macsai, M., & Mojica, G. (2013). Medical Management of Ocular Surface Disease. In E. J. Holland, M. J. Mannis, & W. B. Lee (Eds.), Ocular Surface Disease: Cornea, Conjunctiva and Tear Film (pp. 271-281). W.B. Saunders. https://doi.org/10.1016/B978-1-4557-2876-3.00034-1
- [Background] Mahmoodi AN, Patel P, Kim PY. Ketorolac. 2024 Feb 28. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK545172/ PMID 31424756
- [Background] Shin DH, Frenkel RE, David R, Cheetham JK. Effect of topical anti-inflammatory treatment on the outcome of laser trabeculoplasty. The Fluorometholone-Laser Trabeculoplasty Study Group. Am J Ophthalmol. 1996 Sep;122(3):349-54. doi: 10.1016/s0002-9394(14)72061-6. PMID 8794707
- [Background] Realini T, Charlton J, Hettlinger M. The impact of anti-inflammatory therapy on intraocular pressure reduction following selective laser trabeculoplasty. Ophthalmic Surg Lasers Imaging. 2010 Jan-Feb;41(1):100-3. doi: 10.3928/15428877-20091230-18. PMID 20128578
- [Background] Mermoud A, Pittet N, Herbort CP. Inflammation patterns after laser trabeculoplasty measured with the laser flare meter. Arch Ophthalmol. 1992 Mar;110(3):368-70. doi: 10.1001/archopht.1992.01080150066030. PMID 1543456
- [Background] Herbort CP, Mermoud A, Schnyder C, Pittet N. Anti-inflammatory effect of diclofenac drops after argon laser trabeculoplasty. Arch Ophthalmol. 1993 Apr;111(4):481-3. doi: 10.1001/archopht.1993.01090040073033. PMID 8470978
- [Background] Rebenitsch RL, Brown EN, Binder NR, Jani A, Bonham AJ, Krishna R, Pikey K. Effect of topical loteprednol on intraocular pressure after selective laser trabeculoplasty for open-angle glaucoma. Ophthalmol Ther. 2013 Dec;2(2):113-20. doi: 10.1007/s40123-013-0018-z. Epub 2013 Aug 31. PMID 25135811
- [Background] Kim YY, Glover BK, Shin DH, Lee D, Frenkel RE, Abreu MM. Effect of topical anti-inflammatory treatment on the long-term outcome of laser trabeculoplasty. Fluorometholone-Laser Trabeculoplasty Study Group. Am J Ophthalmol. 1998 Nov;126(5):721-3. doi: 10.1016/s0002-9394(98)00177-9. PMID 9822239
- [Background] Gracner T. Impact of Short-Term Topical Steroid Therapy on Selective Laser Trabeculoplasty Efficacy. J Clin Med. 2021 Sep 19;10(18):4249. doi: 10.3390/jcm10184249. PMID 34575360
- [Background] Dahlgren T, Ayala M, Zetterberg M. The impact of topical NSAID treatment on selective laser trabeculoplasty efficacy. Acta Ophthalmol. 2023 May;101(3):266-276. doi: 10.1111/aos.15276. Epub 2022 Oct 18. PMID 36259097
- [Background] Chen YS, Hung HT, Guo SP, Chang HC. Effects of anti-inflammatory treatment on efficacy of selective laser trabeculoplasty: a systematic review and meta-analysis. Expert Rev Clin Pharmacol. 2021 Dec;14(12):1527-1534. doi: 10.1080/17512433.2021.1981860. Epub 2021 Sep 24. PMID 34524035
- [Background] Jinapriya D, D'Souza M, Hollands H, El-Defrawy SR, Irrcher I, Smallman D, Farmer JP, Cheung J, Urton T, Day A, Sun X, Campbell RJ. Anti-inflammatory therapy after selective laser trabeculoplasty: a randomized, double-masked, placebo-controlled clinical trial. Ophthalmology. 2014 Dec;121(12):2356-61. doi: 10.1016/j.ophtha.2014.07.017. Epub 2014 Sep 16. PMID 25234015
- [Background] De Keyser M, De Belder M, De Groot V. Randomized Prospective Study of the Use of Anti-Inflammatory Drops After Selective Laser Trabeculoplasty. J Glaucoma. 2017 Feb;26(2):e22-e29. doi: 10.1097/IJG.0000000000000522. PMID 27552500
- [Background] Polat J, Grantham L, Mitchell K, Realini T. Repeatability of selective laser trabeculoplasty. Br J Ophthalmol. 2016 Oct;100(10):1437-41. doi: 10.1136/bjophthalmol-2015-307486. Epub 2016 Feb 1. PMID 26834070
- [Background] Avery N, Ang GS, Nicholas S, Wells A. Repeatability of primary selective laser trabeculoplasty in patients with primary open-angle glaucoma. Int Ophthalmol. 2013 Oct;33(5):501-6. doi: 10.1007/s10792-013-9729-3. Epub 2013 Jan 31. PMID 23371484
- [Background] Kramer TR, Noecker RJ. Comparison of the morphologic changes after selective laser trabeculoplasty and argon laser trabeculoplasty in human eye bank eyes. Ophthalmology. 2001 Apr;108(4):773-9. doi: 10.1016/s0161-6420(00)00660-6. PMID 11297496
- [Background] Wong MO, Lee JW, Choy BN, Chan JC, Lai JS. Systematic review and meta-analysis on the efficacy of selective laser trabeculoplasty in open-angle glaucoma. Surv Ophthalmol. 2015 Jan-Feb;60(1):36-50. doi: 10.1016/j.survophthal.2014.06.006. Epub 2014 Jul 2. PMID 25113610
- [Background] Quigley HA. Number of people with glaucoma worldwide. Br J Ophthalmol. 1996 May;80(5):389-93. doi: 10.1136/bjo.80.5.389. PMID 8695555
- [Background] Groth SL, Albeiruti E, Nunez M, Fajardo R, Sharpsten L, Loewen N, Schuman JS, Goldberg JL. SALT Trial: Steroids after Laser Trabeculoplasty: Impact of Short-Term Anti-inflammatory Treatment on Selective Laser Trabeculoplasty Efficacy. Ophthalmology. 2019 Nov;126(11):1511-1516. doi: 10.1016/j.ophtha.2019.05.032. Epub 2019 Jun 6. PMID 31444008
- [Background] Hodge WG, Damji KF, Rock W, Buhrmann R, Bovell AM, Pan Y. Baseline IOP predicts selective laser trabeculoplasty success at 1 year post-treatment: results from a randomised clinical trial. Br J Ophthalmol. 2005 Sep;89(9):1157-60. doi: 10.1136/bjo.2004.062414. PMID 16113372
- [Background] Melamed S, Ben Simon GJ, Levkovitch-Verbin H. Selective laser trabeculoplasty as primary treatment for open-angle glaucoma: a prospective, nonrandomized pilot study. Arch Ophthalmol. 2003 Jul;121(7):957-60. doi: 10.1001/archopht.121.7.957. PMID 12860797
- [Background] Ayala M, Chen E. Comparison of selective laser trabeculoplasty (SLT) in primary open angle glaucoma and pseudoexfoliation glaucoma. Clin Ophthalmol. 2011;5:1469-73. doi: 10.2147/OPTH.S25636. Epub 2011 Oct 12. PMID 22069348
- [Background] Shazly TA, Smith J, Latina MA. Long-term safety and efficacy of selective laser trabeculoplasty as primary therapy for the treatment of pseudoexfoliation glaucoma compared with primary open-angle glaucoma. Clin Ophthalmol. 2010 Dec 16;5:5-10. doi: 10.2147/OPTH.S15952. PMID 21311650
- [Background] Latina MA, Park C. Selective targeting of trabecular meshwork cells: in vitro studies of pulsed and CW laser interactions. Exp Eye Res. 1995 Apr;60(4):359-71. doi: 10.1016/s0014-4835(05)80093-4. PMID 7789416
- [Background] Koucheki B, Hashemi H. Selective laser trabeculoplasty in the treatment of open-angle glaucoma. J Glaucoma. 2012 Jan;21(1):65-70. doi: 10.1097/IJG.0b013e3182027596. PMID 21278588
- [Background] Alon S. Selective Laser Trabeculoplasty: A Clinical Review. J Curr Glaucoma Pract. 2013 May-Aug;7(2):58-65. doi: 10.5005/jp-journals-10008-1139. Epub 2013 May 9. PMID 26997784
- [Background] Rothman, A. L., Delwadia, N. A., Sarwal, R., Stinnett, S. S., Lee, P. P., Herndon, L. W., & Challa, P. (2014). A Comparison of Topical Steroids Versus Non-Steroidal Anti-Inflammatory Drugs after Selective Laser Trabeculoplasty. Investigative Ophthalmology & Visual Science, 55(13), 6158-6158.
- [Background] Park CH, Latina MA, Schuman JS. Developments in laser trabeculoplasty. Ophthalmic Surg Lasers. 2000 Jul-Aug;31(4):315-22. No abstract available. PMID 10928669